CLINICAL TRIAL: NCT01579123
Title: Prospective Trial Comparing Laser Atherectomy to Angioplasty With/Without Stenting for Infrageniculate Peripheral Disease
Brief Title: Laser Atherectomy Versus Angioplasty for the Treatment of Critical Limb Ischemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 012-010
Record Dates: First submitted 2012-04-13; First posted 2012-04-17 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Critical Limb Ischemia
Keywords: Laser atherectomy; Critical Limb Ischemia; Angioplasty
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia | interventions — Angioplasty

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laser atherectomy (Active Comparator)
  Interventions: Procedure: Laser atherectomy
- Angioplasty (Active Comparator)
  Interventions: Procedure: Angioplasty

INTERVENTIONS:
Procedure: Angioplasty — With angioplasty, a catheter is guided to the portion of the artery that is narrowed or blocked off. A balloon that is attached to the end of the catheter will be inflated which dilates or expands the artery in the area where the narrowing or blockage is located. Based on the angiogram and extent of disease, the physician may place a stent (small mesh tube that is used to treat narrow or weak arteries in the body) during the angioplasty.
  Arms: Angioplasty
Procedure: Laser atherectomy — Laser atherectomy uses a catheter that emits high energy light (laser) to unblock the artery. The catheter is moved through the artery until it reaches the blockage. Laser energy is used to essentially vaporize the blockage inside the vessel.
  Arms: Laser atherectomy

SUMMARY:
The reason the investigators are doing this study is to compare the results of laser atherectomy versus angioplasty with or without the placement of a stent in the artery. A stent is a metal tube used to open up narrow arteries in the body.

DETAILED DESCRIPTION:
People with peripheral artery disease that has severely reduced blood flow in their lower leg are usually treated with surgical bypass. This condition is known as Critical Limb Ischemia or CLI. Over the last decade, advances in techniques and tools have allowed surgeons to more aggressively treat complex cases. Studies have shown successful treatment of CLI with endovascular techniques (less invasive surgical procedures through a small incision for the treatment of vascular disease), including laser atherectomy and angioplasty. Surgical guidelines are not clear as to the best procedure to use for CLI. To the best of our knowledge, a study comparing laser atherectomy and angioplasty has not been done. Laser atherectomy works by releasing ultraviolet light which is absorbed by the plaque in the arteries. This will then get rid of the plaque. Angioplasty is a procedure used to open blocked or narrowed arteries. Currently, it is not known if laser atherectomy has better results than angioplasty.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Male or female (non-pregnant females)
* Patients with peripheral artery disease that has progressed to critical limb ischemia (CLI)
* Patients undergoing angiography with possible intervention for Rutherford Class 4-6 limb ischemia that may benefit from revascularization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-02; Primary Completion 2016-09-26 (Actual); Study Completion 2016-09-26 (Actual)

PRIMARY OUTCOMES:
Outcome measure: difference in patency rates | one year

CONTACTS AND LOCATIONS:
Overall Officials: William Shutze, MD, Principal Investigator — Baylor Jack and Jane Hamilton Heart Hospital
Locations (3):
- United States (3):
  - Baylor Jack and Jane Hamilton Heart Hospital, Dallas, Texas
  - Baylor Regional Medical Center at Plano, Plano, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas